CLINICAL TRIAL: NCT04291456
Title: Open-Label Trial of Minocycline in Early Multiple Sclerosis: Confirmation of Treatment Benefit
Brief Title: Minocycline in MS: Confirmation of Benefit
Acronym: MS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Completion is not possible due to recruitment concerns
Sponsor: University of Calgary (Other)
Collaborators: Hotchkiss Brain Institute, University of Calgary (Other); Multiple Sclerosis Society of Canada (Other)
Responsible Party: Principal Investigator, Dr. Luanne Metz, Professor, Department of Clinical Neurosciences, University of Calgary, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MinoMS-2019
Record Dates: First submitted 2019-11-18; First posted 2020-03-02 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome
Keywords: Multiple Sclerosis; Clinically Isolated syndrome; Minocycline
MeSH Terms: conditions — Multiple Sclerosis; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: Non-inferiority Design
Masking Description: A blinded physician will complete the neurologic exam and determine the EDSS (and be blinded as to which trial the patient is participating in) and the radiologists reading the MRI scans will be blinded that the MRI scans are part of a clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minocycline (Experimental): Minocycline 100 mg oral twice daily for up to 24 month
  Interventions: Drug: Minocycline 100mg

INTERVENTIONS:
Drug: Minocycline 100mg — Single-arm trial of minocycline 100 mg twice daily

SUMMARY:
This is an open-label, single-arm clinical trial. Trial participants will include men and women, aged 18-60 years who have had a first demyelinating event within the previous 180 days and who have brain magnetic resonance imaging (MRI) with at least two brain T2 lesions which are at least 3 mm in diameter, and at least one of which is ovoid or periventricular or infra-tentorial. Treatment with minocycline until the endpoint is reached or to a maximum of 24 months or until the last-enrolled participant reaches their 12 month visit.

DETAILED DESCRIPTION:
Background: Multiple sclerosis (MS) is a chronic autoimmune disease of the central nervous system (CNS) characterized by the presence of multifocal lesions with inflammation, demyelination and axonal injury. Most people with MS present with a first clinical demyelinating event. This trial will determine the effects of minocycline treatment after a first clinical demyelinating event.

The investigators recently showed that minocycline, a second-generation tetracycline antibiotic with immune modulating properties, delays conversion from a first clinical demyelinating event to MS within 6 months. While benefit remained significant at 12 months, the investigators were unable to confirm benefit at 24 months. Another trial is needed to confirm the benefit at 6 and 12 months and to determine if the benefit lasts to 24 months. Since this earlier trial the diagnostic criteria for MS have changed and most people with first clinical demyelinating events, previously called a clinically isolated syndrome (CIS), who meet the trial inclusion criteria can now be diagnosed with MS. The outcome of this trial remains clinically important however because it represents the time until new disease activity occurs. It is new activity (brain inflammation or brain damage) which the investigators are trying to prevent with treatment. In Alberta, other proven therapies for CIS, even when MS can now be diagnosed at onset, are not reimbursed by Alberta Blue Cross. Therefore, most people still do not have access to treatment, other than minocycline. Minocycline is therefore a reasonable treatment at this stage of the disease. While the investigators have been lobbying for these reimbursement criteria to be changed there will still be delays in access to other therapies. This will make minocycline valuable, at least as a bridge therapy, while waiting for the option of starting other therapies. Therefore, confirming its' efficacy remains clinically important.

Objective: This proposal will allow the investigators to confirm that minocycline treatment reduces the risk in individuals with a first clinical demyelinating event (CIS or CIS/MS) to have further inflammatory disease activity that is equivalent to the endpoint indicating they converted to MS (by 2005 McDonald MS Criteria).

Patient Population: Participants must meet the same inclusion and exclusion criteria that were used in the investigators previous phase III minocycline trial. These criteria are identical to those of the investigators earlier CIS trial and very similar to other CIS trials. In addition, to assure the cohort remains consistent with participants in previous CIS trials, the investigators will monitor the characteristics of the participating population to assure they reflect the majority of previous CIS trials. The investigators expect the time since onset of CIS may need to be reduced during the trial to ensure the investigators limit the number of participants with longer time from onset to match the investigators earlier trial. This will be monitored closely.

Recruitment: Patients referred to the Calgary MS Clinic with new onset of suspected MS are generally seen within 4 weeks of referral. An MRI scan of their brain will have been completed prior to referral or will be arranged on an urgent basis. This will be the screening/baseline MRI. Patients are routinely assessed for conditions that mimic MS as standard practice in the MS Clinic. If a diagnosis of CIS or CIS/MS is made they are educated about their diagnosis, informed of the risk of MS and of further CNS inflammation (clinical, or subclinical if detected by MRI), and they are offered treatments that may reduce these risks. Clinical and MRI follow-up are arranged and they are advised to contact a clinic nurse if they have new or worsening neurologic symptoms. Current approved therapies for MS are not reimbursed through the Alberta Blue Cross special authorization program until a diagnosis of MS is confirmed and a second inflammatory event has occurred. Therefore, few patients initiate the currently approved MS therapies which cost $13,154 to $34,780 per year. Even a co-pay of 20% is very expensive. However, most patients can afford minocycline 100 mg twice daily (less than $500 per year) and therefore many now choose to start it. Most others choose no treatment. Patients diagnosed with CIS or CIS/MS will be invited to be screened for eligibility to participate in this open-label trial. All consenting patients who meet the study criteria will be enrolled.

Over 48 months, 148 patients will be enrolled. Up to 200 patients may be screened because some screened patients will not meet the MRI criteria for inclusion and some may choose to take another treatment.

Treatment: Study participants will be included in this study if they decide to start treatment with minocycline. Participants who enroll and take at least one dose of minocycline will be evaluated in the intention to treat population. Participants will be asked to continue minocycline and trial participation for up to 24 months but will be discontinued earlier if they reach the study endpoint (MS according to the 2005 McDonald criteria). Continuation of minocycline after this period will be decided by the participant and their neurologist as this period will not be part of the clinical trial.

Participants will be included in a per-protocol analysis group if they take 80% of the prescribed minocycline and have all on study clinical and imaging evaluations prior to reaching the study endpoint. Adherence will be determined based on drug dispensed and pill counts. Participants will be asked to bring in their empty and partially used pill bottles for a pill count. Other MS disease modifying therapies, chronic systemic steroids, and investigational therapies are prohibited. Use of contraception during treatment with minocycline will be required for sexually active participants. Use of other concurrent medications will not be influenced by study participation.

Study Procedures: Clinic visits will occur at screening, baseline, and months 3, 6, 12, 18 and 24, and telephone visits will occur at months 1, 9, 15 and 21. A brief month 1 clinic visit will be required for an EDSS if the participants initial clinical event had not resolved before their screening EDSS. The screening and baseline visit may be on the same day. MRI scans will be done at baseline (or within the previous 2 weeks), and at months 3, 6, 12 and 24 (+/- 14 days). The timing of clinical assessments and MRI scans in the minocycline group will mirror the investigators previous trial which reflected previous CIS trials. Participants will continue in the study until month 24 or until they reach the primary endpoint. They will be considered early drop-outs if they discontinue participation before reaching the primary endpoint. Standard clinical follow-up of CIS and CIS/MS patients generally mirrors this pattern of follow-up.

Clinic visits are routine at months 6, 12 and 24. Study visits at months 1, 3 and 18 are required only for the trial. Telephone visits are only for the trial. Brain MRI is routine at months 6, 12 and 24 and clinic patients who have enhancing lesions on their baseline MRI typically also have a scan at 3 months because they are at very high risk of early new disease activity. Study participants without enhancing lesions on their baseline MRI will therefore have an MRI at 3 months only because they are study participants. These are the only MRI scans being done outside of standard clinical practice.

Masking: Clinical assessments and MRI interpretations will be completed by masked assessors. A masked clinician will complete the neurologic exam and EDSS. While this is a single arm study several trials are ongoing at the investigators centre and the assessor will be masked as to which trial the patient is participating in. The radiologist interpreting the MRI will be masked because they will not know that this is a study MRI.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria have to be met for inclusion of a patient into the study:

* Age between 18 and 60 years inclusive. The lower age limit has been set because the McDonald criteria may not be valid in children and adolescents.15 The upper limit is set because the specificity of the diagnostic criteria is likely reduced in older individuals. Individuals between ages 51-60 must have CSF oligoclonal bands or spinal MRI changes typical of demyelination.
* First focal clinical episode suggestive of demyelinating disease within the previous 180 days (measured from onset of the first symptom to treatment start), based on the appearance of a neurological abnormality, present for at least 24 hours. Objective clinical evidence must be present or documented. Patients will be included irrespective of whether the first clinical demyelinating episode was monosymptomatic (i.e. clinical evidence of a single lesion) or polysymptomatic (i.e. clinical evidence of more than one lesion). The period of 90 days is sufficiently long for case finding and screening procedures and for the patient's decision to participate in the study. In our previous trial the protocol was amended to allow inclusion as late as 180 days after onset, but few participants had onset greater than 90 days before randomization and most CIS trials limited enrolment to within 90 days of onset.
* At least two lesions on the T2-weighted brain* MRI scan with a size of at least 3 mm, at least one of which is ovoid or periventricular or infratentorial. This criterion is required because the presence of MRI abnormalities at the time of the first clinical event affect the probability of developing MS. MRI also increases diagnostic certainty by helping to exclude patients with another etiology (e.g. ischemic or neoplastic causes). MRI eligibility will be determined based on the neuroradiologists clinical report. *One lesion on spinal MRI may substitute for one brain lesion as per the 2005 McDonald Criteria.
* Sexually active women of child-bearing potential must agree to use adequate contraception.
* Written informed consent
* Be a registered Calgary MS Clinic patient
* In addition, participants may be enrolled if, as part of their standard care, they initiated and continued treatment with minocycline 100 mg bid and if, in addition to meeting all the previous inclusion criteria, they: completed all baseline activities after onset of the clinical demyelinating event and before of minocycline initiation, if their baseline MRI was completed within 14 days of minocycline initiation.

Exclusion Criteria:

Patients are to be excluded from enrolment if they display any of the following:

* Any disease other than MS that could better explain the patient's signs and symptoms.
* Any previous clinical event reasonably attributable to acute demyelination, regardless of whether medical attention was obtained.
* They have had two or more MRI scans at least 30 days apart to evaluate the CIS event prior to screening. This will reduce the risk of enrolling participants already monitored for active disease.
* Complete transverse myelitis or bilateral optic neuritis.
* Any patient who reaches the 2005 McDMS endpoint by the time of the baseline assessment. This may be based on the occurrence of a new relapse (onset at least 30 days after onset of CIS) or evidence of dissemination in time on the baseline MRI if a previous brain MRI had already been undertaken at least 30 days after onset of CIS.
* Clinically significant liver, renal, or bone marrow dysfunction.
* Any condition that could interfere with MRI or any other evaluation.
* Known allergy or contraindication to gadolinium-DTPA or tetracyclines including estimated GFR (eGFR) less than 60.
* Concurrent participation in any clinical therapeutic trial.
* Pre-treatment with the following substances prior to study enrolment: IFNß, glatiramer acetate (GA), total lymphoid irradiation, anti-lymphocyte monoclonal antibody treatment [e.g. anti-CD4, anti-CD52 (alemtuzumab), anti-CD20 or B-cell depleting agents (rituximab, ocrelizumab) and anti-VLA4 (natalizumab)], teriflunomide, dimethyl fumarate, fingolimod, cladribine, ocrelizumab, mitoxantrone, cyclophosphamide, azathioprine, cyclosporine A, methotrexate, or any other immunomodulating or immunosuppressive drug including other recombinant or non-recombinant cytokines.
* Use, within the previous 3 months, of any treatment known to be used for experimental MS treatment except minocycline in the case where minocycline was initiated to treat CIS or early MS.
* Any other condition or situation that in the opinion of the investigator would either put the patient at risk of worsening health if enrolled in the trial or

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
proportion of participants diagnosed with multiple sclerosis according to the 2005 McDonald Criteria | 6 months
  The endpoint, Multiple sclerosis, is based on reaching the 2005 diagnostic criteria based on the occurrence of a second relapse or a new or enlarging MRI T2 lesion, or a new gadolinium-enhancing lesion on MRI

SECONDARY OUTCOMES:
Proportion of participants diagnosed with multiple sclerosis according to the 2005 McDonald Criteria | 3,6, 12 and 24 months
  The endpoint, Multiple sclerosis, is defined as meeting the 2005 diagnostic criteria for MS which is based on the occurrence of a second relapse or a new or enlarging MRI T2 lesion, or a new gadolinium-enhancing lesion on MRI AND meeting the criteria for dissemination in space based on neurologic exam or MRI lesion distribution, as defined for the published criteria.
The proportion of participants with no evidence of disease activity (NEDA) | 3,6,12,and 24 months
  NEDA is defined as absence of relapse, and absence of any new or enlarging T2 MRI lesions and absence of any enhancing MRI lesions and absence of worsening of disability defined as a change of 1.5 points on the extended disability status scale (EDSS).

CONTACTS AND LOCATIONS:
Overall Officials: Luanne Metz, MD,FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Calgary MS Clinic at Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No